CLINICAL TRIAL: NCT02782754
Title: Treatment of Intracranial Germinoma With Chemotherapy Prior to Reduced Dose and Volume of Radiotherapy
Brief Title: Chemotherapy Plus Reduced Radiotherapy in Intracranial Germinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-10-101
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Intracranial Germinoma
MeSH Terms: conditions — Germinoma | interventions — Carboplatin; Etoposide; Cyclophosphamide; Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intracranial germinoma (Experimental): 1. Four cycles of chemotherapy with carboplatin, etoposide, (+ bleomycin) and cyclophosphamide, etoposide, (+ bleomycin) regimen
  2. Reduced dose of radiotherapy
     * Without seeding: 18 Gy to ventricle + 12.6 Gy to primary site
     * With seeding: craniospinal irradiation 18 Gy + 12.6 Gy to primary site
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Bleomycin; Radiation: Reduced dose of radiotherapy

INTERVENTIONS:
Drug: Carboplatin
Drug: Etoposide
Drug: Cyclophosphamide
Drug: Bleomycin
Radiation: Reduced dose of radiotherapy

SUMMARY:
The purpose of this study is to evaluate the outcome of intracranial germinoma treated with chemotherapy plus reduced radiotherapy.

DETAILED DESCRIPTION:
Treatment outcome of intracranial germinoma is excellent with radiotherapy/chemotherapy. However, late sequelae are unavoidable especially with craniospinal irradiation, and various efforts have been done to reduce the dose and extent of radiotherapy. In this study, chemotherapy and further reduced dose of radiotherapy will be used to minimize the late sequelae in the patients with intracranial germinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven intracranial germinoma

Exclusion Criteria:

* Elevated serum/cerebrospinal fluid alpha-feto protein
* Patients with organ dysfunction as follows (creatinine elevation, ejection fraction, liver function test > CTCAE grade 2)

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Rate of late sequelae | Up to 5 years

SECONDARY OUTCOMES:
Rate of event free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee JW, Lim DH, Sung KW, Cho HW, Ju HY, Yoo KH, Koo HH, Kim JH, Suh YL, Shin HJ. Induction Chemotherapy Reduces Radiation Therapy Dose and Volume in the Treatment of Intracranial Germinoma: Results of the SMC-G13 Trial. Int J Radiat Oncol Biol Phys. 2020 Nov 1;108(3):649-656. doi: 10.1016/j.ijrobp.2020.05.051. Epub 2020 Jun 2. PMID 32502506